CLINICAL TRIAL: NCT03870958
Title: Cost-effectiveness of the Application of Glass Ionomer Cement Sealant (GC Fuji TRIAGE®) in the Prevention of Post-eruptive Fractures in Molars Affected by Molar-Incisor Hipomineralisation: Controlled and Randomized Clinical Trial
Brief Title: Glass Ionomer Cement Sealant in the Prevention of Post-eruptive Fractures in Molars Affected by MIH
Acronym: MIHMex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Isabel Cristina Olegário da Costa (Other)
Collaborators: University of Guadalajara (Other); University of Dublin, Trinity College (Other); Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Sponsor-Investigator, Isabel Cristina Olegário da Costa, PhD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MIHMex
Record Dates: First submitted 2018-12-03; First posted 2019-03-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: This two-arm, parallel group, patient-randomized controlled, superiority trial will have treatment provided in schools. Schoolchildren (age 6-9), presenting at least one MIH molar (n molars = 195,) will have random allocation to treatment with or without the application of a GIC sealant (GC Fuji TRIAGE®, GC Europe, Leuven, Belgium).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GIC sealant (GC Fuji TRIAGE®) (Experimental): Children allocated to this group will receive the same dietary advices and brushing instructions. Additionally, all MIH molars from will receive a GIC sealant (GC Fuji TRIAGE®, GC Europe, Leuven, Belgium).
  Interventions: Procedure: GIC sealant (GC Fuji TRIAGE®)
- Control (Active Comparator): Children allocated to this group will receive the same dietary advices and brushing instructions described in the control arm.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: GIC sealant (GC Fuji TRIAGE®) — Children allocated to this group will receive the same dietary advices and brushing instructions. Additionally, all MIH molars from will receive a GIC sealant (GC Fuji TRIAGE®, GC Europe, Leuven, Belgium).
  Arms: GIC sealant (GC Fuji TRIAGE®)
Procedure: Control — Children allocated to this group will receive the same dietary advices and brushing instructions.
  Arms: Control

SUMMARY:
This trial will compare the application of Glass Ionomer Cement (GIC) sealant with no-intervention for the most clinically- and cost-effective strategy for managing MIH molars without post-eruptive breakdown, in a school setting, using low-technology and child-friendly dental techniques. Methods/Design: This two-arm, parallel group, patient-randomized controlled, superiority trial will have treatment provided in schools. Schoolchildren (age 6-9), presenting at least one MIH molar (n molars = 195,) will have random allocation to treatment with or without the application of a GIC sealant (GC Fuji TRIAGE®, GC Europe, Leuven, Belgium). Baseline measures and outcome data will be assessed through participant report and clinical examination. The primary outcome is the presence of post-eruptive fracture and development of caries lesions. Secondary outcomes are: (1) self-reported dental hypersensitivity; (2) oral health-related-quality of life, reported by children; (3) plaque index, (4) gingival health, (5) caries status (according to ICCMS scores) in primary and permanent teeth; (6) the incremental cost-effectiveness. A trained and calibrated examiner will evaluate the treated teeth every six months post treatment for a period of 36 months. Kaplan-Meier and Cox regression tests will be used to investigate the primary outcome. The Logistic Regression and Poisson Regression Analysis will be used to analyze the secondary outcomes (α=5%).

DETAILED DESCRIPTION:
Background: Molar-Incisor Hypomineralisation (MIH) is defined as a qualitative defect that occurs during the mineralization phase of enamel of at least one first permanent molar. The opacities vary in size and color and are demarcated by healthy enamel. MIH molars present lower mechanical properties when compared to non-affected molars, due to the enamel's decreased mineralization. Allied to that, patients often report dental hypersensitivity, which impairs the mechanical removal of dental plaque; therefore, those molars are more prone to post-eruptive fractures and present higher risk of developing dental caries. This trial will compare the application of Glass Ionomer Cement (GIC) sealant with no-intervention for the most clinically- and cost-effective strategy for managing MIH molars without post-eruptive breakdown, in a school setting, using low-technology and child-friendly dental techniques. Methods/Design: This two-arm, parallel group, patient-randomized controlled, superiority trial will have treatment provided in schools. Schoolchildren (age 6-9), presenting at least one MIH molar (n molars = 195,) will have random allocation to treatment with or without the application of a GIC sealant (GC Fuji TRIAGE®, GC Europe, Leuven, Belgium). Baseline measures and outcome data will be assessed through participant report and clinical examination. The primary outcome is the presence of post-eruptive fracture and development of caries lesions. Secondary outcomes are: (1) self-reported dental hypersensitivity; (2) oral health-related-quality of life, reported by children; (3) plaque index, (4) gingival health, (5) caries status (according to ICCMS scores) in primary and permanent teeth; (6) the incremental cost-effectiveness. A trained and calibrated examiner will evaluate the treated teeth every six months post treatment for a period of 36 months. Kaplan-Meier and Cox regression tests will be used to investigate the primary outcome. The Logistic Regression and Poisson Regression Analysis will be used to analyze the secondary outcomes (α=5%).

ELIGIBILITY:
Inclusion criteria:

* children whose parents or legal guardians accept and sign the informed consent form; -children who assent to participate into the research;
* aged between 6 and 9 years;
* exhibiting good general health conditions and cooperative behavior;
* presenting at least one MIH molar.

Exclusion criteria:

* children presenting health conditions that impair the dental treatment, or children undergoing orthodontic treatment;
* MIH molars that present opacities not located on the occlusal surface, with post-eruptive breakdown, with the occlusal surface totally or partial covered by a gingival operculum, with caries dentine lesion (ICCMS score C), restorations or sealants.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Post-eruptive breakdown | After 12 months
  A "success" will be accounted in cases when the no post-eruptive breakdown is detected, while a "failure" will be considered when a post-eruptive breakdown, atypical restoration, atypical caries or tooth missing due to MIH is perceived.
  Method: clinical evaluation by a calibrated examiner

SECONDARY OUTCOMES:
Caries lesions assessment | Every 6 months up to 36 months
  The dental caries index ICCMS (Ismail et al., 2015) will be used. For that, a visual-tactile exam will be performed with the aid of an OMS probe.
  Method: clinical evaluation by a calibrated examiner
Sealant retention | Every 12 months up to 36 months
  The sealants 'retention will be clinically evaluated and scored as: 0- fully retained sealant; 1- partially retained sealant and 2- sealant absent (Oba et al., 2009). (Hilgert LA et al., 2017)
  Method: clinical evaluation by a calibrated examiner
Oral health-related quality of life (OHRQoL) | Baseline and every 12 months up to 36 months
  All children will be interviewed concerning their OHQoL by a local dentist. For that, the Child Perceptions Questionnaire (CPQ) will be used. This questionnaire has already been adapted and validated into Spanish-language (Carmen Aguilar-Díaz F et al., 2011).
Cost-efficacy of treatments | Baseline, after treatment and every 12 months up to 36 months
  The cost-effectiveness analysis will take into account the direct and indirect costs of the procedures. The time spent in each session will be considered, with the total time spent timed by an external assistant. The numbers of consultations attended to each participant and the procedures performed will be registered.
Hypersensitivity | hypersensitivity will be evaluated at 6-month intervals so that evaluations will be completed in 6, 12, 18, 24, 30 and 36 months by the same examiner.
  A questionnaire will be used which will be applied to children with specific questions, a) presence of hypersensitivity when ingesting hot and cold drinks; b) hypersensitivity when brushing teeth. Clinically it will be used the methodology used by Mehta D, et al., 2015. A cold air stimulus (2-s air blast, approximately 40 psi, from a dental syringe directed perpendicular to the molar surface at 0.5 cm distance). Neighboring teeth were shielded with cotton rolls or with the fingers of the examiner. Immediately after stimulation patients were asked to point to the g visual analog scale VAS scale (no pain = 0 and worst pain = 10 cm) to the nearest full centimeter number describing their pain perception. Brushing the child's teeth will identify if the child has hypersensitivity and the VAS is used in the same way.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Hesse, Professor, Study Chair — Academic Centre for Dentistry in Amsterdam; Isaac M Pedroza Uribe, MSc, Principal Investigator — University of Guadalajara
Locations (1):
- Isaac Murisi Pedroza, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghanim A, Marino R, Manton DJ. Validity and reproducibility testing of the Molar Incisor Hypomineralisation (MIH) Index. Int J Paediatr Dent. 2019 Jan;29(1):6-13. doi: 10.1111/ipd.12433. Epub 2018 Oct 22. PMID 30350324
- [Background] Folayan MO, Chukwumah NM, Popoola BO, Temilola DO, Onyejaka NK, Oyedele TA, Lawal FB. Developmental defects of the enamel and its impact on the oral health quality of life of children resident in Southwest Nigeria. BMC Oral Health. 2018 Sep 27;18(1):160. doi: 10.1186/s12903-018-0622-3. PMID 30261858
- [Background] Ebel M, Bekes K, Klode C, Hirsch C. The severity and degree of hypomineralisation in teeth and its influence on oral hygiene and caries prevalence in children. Int J Paediatr Dent. 2018 Nov;28(6):648-657. doi: 10.1111/ipd.12425. Epub 2018 Sep 23. PMID 30246468
- [Background] Velandia LM, Alvarez LV, Mejia LP, Rodriguez MJ. Oral health-related quality of life in Colombian children with Molar-Incisor Hypomineralization. Acta Odontol Latinoam. 2018 Jun;31(1):38-44. PMID 30056465
- [Background] Fragelli CMB, Souza JF, Bussaneli DG, Jeremias F, Santos-Pinto LD, Cordeiro RCL. Survival of sealants in molars affected by molar-incisor hypomineralization: 18-month follow-up. Braz Oral Res. 2017 Apr 27;31:e30. doi: 10.1590/1807-3107BOR-2017.vol31.0030. PMID 28489117
- [Derived] Schraverus MS, Olegario IC, Bonifacio CC, Gonzalez APR, Pedroza M, Hesse D. Glass Ionomer Sealants Can Prevent Dental Caries but Cannot Prevent Posteruptive Breakdown on Molars Affected by Molar Incisor Hypomineralization: One-Year Results of a Randomized Clinical Trial. Caries Res. 2021;55(4):301-309. doi: 10.1159/000516266. Epub 2021 Jun 9. PMID 34107492